CLINICAL TRIAL: NCT02787304
Title: A Phase 2 Double-blind, Randomized, Placebo-controlled, Dose-finding Study to Evaluate the Safety, Tolerability and Efficacy of Volixibat Potassium, an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi) in Adults With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Volixibat (SHP626) in the Treatment of Adults With Nonalcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP626-201; 2016-000203-82 (EudraCT Number)
Record Dates: First submitted 2016-05-11; First posted 2016-06-01 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: NAFLD activity score; ASBTi; MRI PDFF; NAS; NAFLD; liver disease; ASBT; MRI proton density fat fraction; nonalcoholic steatohepatitis; apical sodium dependent bile acid transporter inhibitor; fatty liver; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver | interventions — volixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SHP626 5 Milligram (mg) (Experimental): Subject will be administered 5 mg SHP626 capsule by orally once daily in a double-blinded fashion
  Interventions: Drug: SHP626
- SHP626 10 Milligram (mg) (Experimental): Subject will be administered 10 mg SHP626 capsule by orally once daily in a double-blinded fashion
  Interventions: Drug: SHP626
- SHP626 20 Milligram (mg) (Experimental): Subject will be administered 20 mg SHP626 capsule by orally once daily in a double-blinded fashion
  Interventions: Drug: SHP626
- Placebo (PBO) (Placebo Comparator): Subject will be administered SHP626 matching PBO capsule by orally once daily in a double-blinded fashion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP626 — 5 mg, 10 mg, and 20 mg of SHP626 capsule by orally once daily in a double-blinded fashion
  Other Names: Volixibat (SHP626)
  Arms: SHP626 10 Milligram (mg); SHP626 20 Milligram (mg); SHP626 5 Milligram (mg)
Drug: Placebo — Matching placebo
  Arms: Placebo (PBO)

SUMMARY:
The purpose of this study is to determine if the investigational treatment volixibat (SHP626) is safe, tolerable and effective in adults with nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

1. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
2. Ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative, as applicable) informed consent to participate in the study.
3. Age 18-80 years inclusive. This inclusion criterion will only be assessed at the first screening visit.
4. Male, or non-pregnant, non-lactating female, who is sexually active and who agrees to comply with the contraceptive requirements of the protocol, or females of non-childbearing potential. Males and females of child-bearing potential who are sexually active must agree to use acceptable contraception during the study and for 30 days following the last dose of the investigational product (IP).
5. Presence of greater than equals to (>=) 5 percent (%) steatosis on screening magnetic resonance imaging (MRI) from a centrally read radiologist performed either during the screening period or within 6 months prior to the first visit.
6. Histologic confirmation of nonalcoholic steatohepatitis (NASH) without cirrhosis (F0-F3) from a centrally read liver biopsy performed either during the screening period or within 6 months prior to the first visit with a NAS of >=4 with a score of at least 1 in each component (steatosis, lobular inflammation, and hepatocyte ballooning).

Exclusion Criteria:

1. Presence of or history of cirrhosis or evidence of decompensated liver disease (example: ascites, variceal bleeding, etc.) or hepatocellular carcinoma.
2. History or presence of other concomitant liver disease as assessed by the investigator or determined by laboratory findings including, but not limited to: active hepatitis B virus (HBV) infection (hepatitis B surface antigen [HBsAg] positive and/or hepatitis B virus deoxyribonucleic acid (HBVDNA) positive; subjects who are hepatitis B core antibody [HBcAb] positive may be eligible as long as HBsAg is negative and HBVDNA is non detectable), active hepatitis C virus (HCV) infection (prior exposure to HCV [defined as HCVAb positive] without a current or prior history of a detectable HCVRNA) may be eligible, alcoholic liver disease, proven autoimmune hepatitis, primary biliary cirrhosis (PBC), primary sclerosing cholangitis (PSC), hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, bile duct obstruction, liver primary or metastatic cancer.
3. Current or recurrent disease that could affect the action, absorption, disposition, or laboratory assessment of the IP (including bile salt metabolism in the intestine) example (e.g,) uncontrolled inflammatory bowel disease, uncontrolled celiac disease, gastric bypass procedures (gastric lap band or gastric sleeve is acceptable), ileal or ileocecal resection, uncontrolled irritable bowel syndrome with predominant diarrhea, or history of chronic diarrhea or loose stools of any etiology.
4. Weight change >=5% after qualifying liver biopsy and/or MRI performed. If the subject had a liver biopsy and/or MRI within 6 months of screening, but experienced a weight change of >=5% since the date of liver biopsy and/or MRI, the liver biopsy and/or MRI must be repeated at screening.
5. Contraindications to MRI (e.g, claustrophobia, coronary stents, coronary implantable devices, girth, etc.). Stents or other devices may be allowed, at the investigator's discretion, if they do not interfere with the functioning of the MRI machine.
6. Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to complete the study.
7. Treatment with Vitamin E, thiazolidinediones (TZD), or glucagon-like peptide-1 receptor agonists (GLP-1 RA) unless subject on a stable dose for 6 months prior to qualifying liver biopsy and not initiated after qualifying liver biopsy and will continue the same dosing regimen throughout study participation.
8. Uncontrolled diabetes defined as HbA1c of >=9.5% within 60 days prior to enrollment.
9. Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) that could affect the action, absorption, or disposition of the IP, or clinical or laboratory assessment. (Current use is defined as use within 14 days of screening). Subjects currently taking insulin will not be excluded; however, they must be on a stable dose for at least 30 days prior to screening, or a sliding scale of insulin is allowed as long as the subject's HbA1c remains less than (<) 9.5%.
10. Use of drugs, herbs or supplements historically associated with causing or worsening NAFLD/NASH for less than 6 months prior to liver biopsy, or initiated any time after liver biopsy performed, including the use of total parenteral nutrition (TPN).
11. Serum aspartate aminotransferase (AST) greater than (>) 7 times upper limit of normal (ULN) at screening.
12. Serum alanine aminotransferase (ALT) >7 times ULN at screening.
13. Elevated serum creatinine >=2.0 milligram/deciliter (mg/dL).
14. International normalized ratio (INR) >1.3
15. Total bilirubin (TB) >2.0 times ULN at screening (Except for documented Gilbert's syndrome with bilirubin levels 20 micromole per liter (mcmol/L) to 90 mcmol/L (1.2 to 5.3 mg/dL) and with a ratio of unconjugated/conjugated bilirubin that is commensurately higher).
16. Platelet count <130 × 10^9/liter (L)
17. Medical history of impaired hemostasis or use of anticoagulant medication (use of antiplatelet medications, such as low-dose, that is 81 mg, aspirin [ASA] or clopidogrel [Plavix] will be allowed).
18. Uncontrolled thyroid disease.
19. Type 1 diabetes mellitus.
20. Known or suspected intolerance or hypersensitivity to the IP, closely-related compounds, or any of the stated ingredients.
21. Known history of alcohol or other substance abuse within the last year or at any time during the study based on investigator's discretion. Weekly alcohol intake greater than 21 grams/day for males and 14 grams/day for females on average or inability to reliably quantify alcohol consumption based on investigator's judgment.
22. Within 6 months of MRI and liver biopsy:

    * Have used any IP.
    * Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.
23. Inability to safely obtain a liver biopsy.
24. Females who are pregnant, planning to become pregnant, or are breastfeeding, or males who are planning to father a child during study participation.
25. The anticipated need for a surgical procedure during the study that could interfere with the treatment.
26. Known positivity for human immunodeficiency virus (HIV) infection.
27. Cancer within 5 years of screening, except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma that has been treated with no evidence of recurrence.
28. History of noncompliance with medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to noncompliance with the study protocol.
29. Any other conditions or abnormalities which, in the opinion of the investigator, may compromise the safety of the subject, or interfere with the subject participating.
30. Subject is currently enrolled in this study at any study site (unless the subject is transferring to another qualified study site with prior sponsor approval).
31. Subjects who are employees at the unit of the investigational site that is conducting the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (65):
- United States (49):
  - Southern California Research Center, Coronado, California
  - Fresno Clinical Research Center, Fresno, California
  - Ceders-Sinai Medical Center, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - George Washington (GW) Medical Faculty Associates, Washington D.C., District of Columbia
  - Schiff Center for Liver Diseases, Miami, Florida
  - South Florida Center of Gastroenterology, Wellington, Florida
  - Internal Medicine Associates of Wellstar Atlanta Medical, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - The Queen's Medical Center - Liver Center, Honolulu, Hawaii
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Liver Research Center, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, Catonsville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health Inc., Manhasset, New York
  - Concorde Medical Group PLLC, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Center for Liver Disease, Charlotte, North Carolina
  - DUMC-Gastroenterology, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Carolinas Center for Liver Disease, Statesville, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinsearch, LLC, Chattanooga, Tennessee
  - University of TN Health Science Center, Memphis, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - Methodist Health Systems Clinical, Dallas, Texas
  - Baylor College of Medicine - Advanced Liver Therapies, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - DHAT Research Institute, Richardson, Texas
  - UVM Medical Center, Burlington, Vermont
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - UW Digestive Health Center (DHC), Madison, Wisconsin
- Canada (6):
  - University of Calgary Liver Unit, Calgary, Alberta
  - LAIR Centre, Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Nova Scotia Heath Authority, Halifax, Nova Scotia
  - Toronto Liver Centre, Toronto, Ontario
  - CRCHUM, Montreal, Quebec
- UPR: Medical Sciences Campus, San Juan, Puerto Rico
- United Kingdom (9):
  - Royal Free Hospital, Hampstead, London
  - Norfolk & Norwich University Hospital, Norwich, Norfolk
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - NHS Tayside, Dundee, Tayside
  - University Hospital Birmingham, Birmingham, West Midlands
  - Royal London Hospital, London
  - Nottingham Digestive Diseases Centre and Biomedical Research Unit, Nottingham
  - Abertawe Bro Morgannwg University, Swansea
  - York Clinical Research Facility, York

REFERENCES:
- [Derived] Newsome PN, Palmer M, Freilich B, Sheikh MY, Sheikh A, Sarles H, Herring R, Mantry P, Kayali Z, Hassanein T, Lee HM, Aithal GP; Volixibat in Adults study group. Volixibat in adults with non-alcoholic steatohepatitis: 24-week interim analysis from a randomized, phase II study. J Hepatol. 2020 Aug;73(2):231-240. doi: 10.1016/j.jhep.2020.03.024. Epub 2020 Mar 29. PMID 32234329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Started | 49 | 50 (One subject was randomized and received 1 dose of study drug but withdrew from the study.) | 49 | 49
Completed | 13 | 12 | 8 | 15
Not Completed | 36 | 38 | 41 | 34
Not completed — Adverse Event | 9 | 3 | 8 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Noncompliance with study drug | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 25 | 31 | 31 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO) | Total
Number analyzed (Participants) | 49 | 49 | 49 | 49 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated as the difference between date of birth and date of informed consent, rounded down to the last whole year.
  years | 52.8 (14.13) | 53.0 (11.84) | 53.2 (13.61) | 53.4 (11.75) | 53.1 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 25 | 32 | 118
  Male | 22 | 15 | 24 | 17 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 7 | 7 | 33
  Not Hispanic or Latino | 40 | 39 | 42 | 42 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 4 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 4 | 4 | 9
  White | 46 | 47 | 41 | 41 | 175
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Binary Response on Liver Histology Between Volixibat (SHP626) and Placebo at Week 48
Description: Binary response indicating (yes/no) whether a subject responded at week 48 with a reduction of at least 2 points, without worsening of fibrosis, from baseline nonalcoholic fatty liver disease (NAFLD) activity score (NAS). The NAS grades NAFLD on liver biopsy based on the individual scoring of steatosis, inflammation and ballooning. The NAS is assessed on a scale of 0 to 8 with higher scores indicating more severe disease and lower scores indicating less severe disease. NAS is obtained by adding steatosis(assessed on a scale of 0 to 3), inflammation (assessed on a scale of 0 to 3) and ballooning (assessed on a scale of 0 to 2).
Time Frame: Baseline, Week 48
Population: Full Analysis Set for subjects with liver biopsy at both Baseline and Week 48 (post hoc analysis) at the time of the interim analysis
Measure: Count of Participants; unit: Participants
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 11 | 11 | 8 | 13
Participants | 4 | 2 | 3 | 5

2. Secondary Outcome: Change From Baseline to Week 48 on Liver Histology
Description: Change in liver histology will be measured by the individual NAS components (ballooning, inflammation, steatosis). The NAS grades NAFLD on liver biopsy based on the individual scoring of steatosis, inflammation and ballooning. The NAS is assessed on a scale of 0 to 8 with higher scores indicating more severe disease and lower scores indicating less severe disease. NAS is obtained by adding steatosis (assessed on a scale of 0 to 3), inflammation (assessed on a scale of 0 to 3) and ballooning (assessed on a scale of 0 to 2).
Time Frame: Baseline, Week 48
Population: Safety Analysis Set for subjects with liver biopsy at both Baseline and Week 48 (post hoc analysis) at the time of the interim analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 11 | 11 | 8 | 13
score on a scale
  NAS - steatosis | -0.5 (0.82) | -0.2 (0.87) | -0.5 (0.93) | -0.3 (0.85)
  NAS - ballooning | -0.3 (0.9) | -0.2 (0.75) | 0.0 (0.93) | -0.7 (0.85)
  NAS - inflammation | -0.2 (0.75) | -0.5 (0.93) | -0.5 (0.76) | -0.7 (0.95)

3. Secondary Outcome: Change From Baseline to Week 48 on Hepatic Steatosis
Description: Change in hepatic steatosis will be evaluated by measuring the reduction of liver fat with magnetic resonance imaging-proton density fat-fraction (MRI-PDFF) and stratified by treatment group.
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis
Measure: Mean (Standard Deviation); unit: absolute percentage
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 13 | 12 | 8 | 13
absolute percentage | -2.68 (4.801) | -1.31 (7.555) | -3.89 (4.474) | -1.34 (5.478)

4. Secondary Outcome: Change From Baseline to Week 48 on Liver Histology
Description: Change in liver histology will be measured by fibrosis stage. Fibrosis stage is assessed on a scale of 0-4 with higher scores indicating more severe disease and lower scores indicating less severe disease (F0 = no fibrosis, F4 = cirrhosis).
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 11 | 11 | 8 | 13
units on a scale
  Fibrosis Score Baseline | 1.8 (1.08) | 2.2 (0.98) | 1.5 (1.07) | 1.4 (0.96)
  Fibrosis Score Week 48 | 1.5 (1.13) | 2.2 (1.25) | 2.1 (1.25) | 1.3 (0.95)

5. Secondary Outcome: Number of Participants With Resolution of NASH at Week 48
Description: Resolution of NASH is defined as total absence of ballooning [score = 0], absent or mild inflammation [score 0-1], steatosis can be present [score 0-3]) without worsening of fibrosis as assessed by liver histology at Week 48.
Time Frame: Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 11 | 11 | 8 | 13
Participants | 2 | 3 | 2 | 5

6. Secondary Outcome: Change From Baseline to Week 48 on Serum Liver-related Biochemistry
Description: Serum liver-related biochemistry will be analysed by measuring alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and gamma glutamyl transferase (GGT).
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 18 | 16 | 15 | 20
U/L
  ALT change from Baseline | 1.2 (25.83) | 4.2 (33.65) | -6.9 (37.91) | -0.2 (24.93)
  AST change from Baseline | 7.6 (16.57) | 10.6 (31.23) | -7.2 (27.08) | -0.8 (14.45)
  ALP change from Baseline | 5.3 (9.62) | -0.9 (27.37) | -0.1 (14.82) | -0.7 (10.66)
  GGT change from Baseline | 8.8 (46.24) | 5.2 (47.24) | -8.8 (45.43) | -8.5 (41.11)

7. Secondary Outcome: Change From Baseline to Week 48 on Serum Liver-related Biochemistry
Description: Serum liver-related biochemistry will be analysed by measuring total bilirubin (TB).
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 18 | 16 | 15 | 20
mg/dL | 0.019 (0.2198) | 0.124 (0.2872) | 0.060 (0.2730) | 0.058 (0.1762)

8. Secondary Outcome: Change From Baseline to Week 48 on Metabolic Indicators
Description: Metabolic indicators will be assessed by measuring fasting serum glucose levels and insulin levels.
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis. For insulin levels, samples were collected but due to study termination for futility after the interim analysis, an analysis of this outcome measure was not performed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 18 | 16 | 15 | 20
mg/dL | 3.5 (40.07) | -5.0 (23.11) | 1.6 (21.31) | 15.6 (45.84)

9. Secondary Outcome: Change From Baseline to Week 48 on Metabolic Indicators
Description: Metabolic indicators will be assessed by measuring hemoglobin A1c (HbA1c).
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis.
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 18 | 16 | 15 | 20
percentage of glycated hemoglobin | -0.0003 (0.00559) | -0.0008 (0.00552) | -0.0020 (0.00426) | 0.0033 (0.00701)

10. Secondary Outcome: Change From Baseline to Week 48 on Serum Lipids
Description: Serum lipids level will be measured by calculating fasting total cholesterol, high-density lipoprotein-cholesterol (HDL-C), low-density lipoprotein-cholesterol (LDL-C), and triglycerides.
Time Frame: Baseline, Week 48
Population: Safety Analysis Set (post hoc analysis) - for subjects with Week 48 data at the time of interim analysis
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
Number analyzed (Participants) | 18 | 16 | 15 | 20
mg/dL
  Fasting total cholesterol change from Baseline | -13.4 (32.06) | -19.1 (38.26) | -7.6 (26.94) | 4.7 (30.38)
  HDL-C change from Baseline | 1.8 (6.72) | 2.2 (10.36) | 2.7 (6.56) | 0.0 (6.74)
  LDL-C change from Baseline | -13.4 (27.38) | -19.5 (31.78) | -9.0 (22.37) | -0.8 (26.12)
  Triglycerides change from Baseline | -9.5 (37.05) | -0.2 (92.34) | -7.2 (71.62) | 28.7 (52.48)

ADVERSE EVENTS:
Time Frame: Up to Visit 10 (Week 52)
Arm/Group | SHP626 5 Milligram (mg) | SHP626 10 Milligram (mg) | SHP626 20 Milligram (mg) | Placebo (PBO)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/49 | 0/49 | 1/49
Other Adverse Events (participants affected / at risk) | 44/49 | 44/49 | 42/49 | 37/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP626 5 Milligram (mg) (N=49) | SHP626 10 Milligram (mg) (N=49) | SHP626 20 Milligram (mg) (N=49) | Placebo (PBO) (N=49)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP626 5 Milligram (mg) (N=49) | SHP626 10 Milligram (mg) (N=49) | SHP626 20 Milligram (mg) (N=49) | Placebo (PBO) (N=49)
Diarrhoea (Gastrointestinal disorders) | 38 (43) | 35 (46) | 35 (47) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 9 (10) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (6) | 4 (6) | 7 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (2) | 7 (8) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 2 (5)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 1 (1) | 3 (4) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (4) | 3 (3) | 3 (3) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (1) | 3 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
At the Week 24 Interim Analysis, no differences were observed between any dose of Volixibat and placebo based on absolute change in steatosis from baseline, as assessed by MRI hepatic PDFF, and % change from baseline in ALT; the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT02787304/SAP_000.pdf
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT02787304/Prot_001.pdf